CLINICAL TRIAL: NCT05845775
Title: Evaluation Of The Effect Of Morphological Structure On Dilatational Tracheostomy Interference Location And Complications By Ultrasonography And Fiberoptic Bronchoscopy
Brief Title: Evaluation Of The Effect Of Morphological Structure On Dilatational Tracheostomy Interference Location And Complications
Status: Completed | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, MD, Clinical Professor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Akdeniz University Medicine
Record Dates: First submitted 2023-04-15; First posted 2023-05-06 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Tracheostomy Complication
Keywords: Complications; Intensive care unit; Tracheostomy
MeSH Terms: interventions — Bronchoscopy; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- percutaneous dilatational tracheostomy: Patients assigned to percutaneous dilatational tracheostomy
  Interventions: Procedure: Percutaneous dilatational tracheostomy; Device: Bronchoscopy; Device: ultrasonography; Diagnostic Test: Bronchoscopy application; Diagnostic Test: Ultrasound examination

INTERVENTIONS:
Procedure: Percutaneous dilatational tracheostomy — The percutaneous dilatational tracheostomy procedure will be performed via fiberoptic bronchoscopy
Device: Bronchoscopy — Fiberoptic bronchoscopy
Device: ultrasonography — ultrasonography
Diagnostic Test: Bronchoscopy application — Fiberoptic bronchoscopy application
Diagnostic Test: Ultrasound examination — Ultrasound examination

SUMMARY:
In recent years, percutaneous dilatational tracheostomy has become a frequently performed procedure in intensive care units. However, tracheostomy procedure has risks of complications of varying severity, such as bleeding, subcutaneous emphysema, posterior tracheal wall damage, tracheal stenosis, infection, and fistula in the early and late periods. It is important to determine the anatomical position for tracheal puncture in reducing the risk of complications. It is not always possible to determine the optimal anatomical position for tracheal puncture in patients in the intensive care unit due to reasons such as obesity patient positioning difficulties and tracheal deviation. In this stuy, we have purpose to evaluate the effect of the morphological structure of patients on the dilatational tracheostomy interference location and complications in the percutaneous dilatational tracheostomy procedure (using anatomical landmarks) performed with the forceps dilatation technique, using fiberoptic bronchoscopy and ultrasonography.

DETAILED DESCRIPTION:
A prospective observational study will be conducted in the Akdeniz University Hospital at the department of Anesthesiology and Intensive Care. Tracheostomy incision site will be determined by using anatomical landmark in all patients. Before the procedure, detailed anatomical measurements showing the morphological structure of the patient (neck thickness, thyromental distance, thyroid cartilage measurement, cricoid cartilage measurement, jugulomental distance, distance between clavicle and cricoid cartilage) will be recorded. In addition, measurements will be made and recorded by ultrasonography. In all patients, the percutaneous dilatational tracheostomy procedure will be performed via fiberoptic bronchoscopy and the tracheal puncture level will be confirmed. Tracheostomy related complications will also be recorded.

ELIGIBILITY:
Example:

● Patients undergoing percutaneous dilatational tracheotomy

Inclusion Criteria:

● Clinical indication for tracheostomy

Exclusion Criteria:

* Age <18
* Patients with severe coagulopathy
* Unsuitable anatomy (e.g., previous cervical surgery, cervical trauma, or tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were decided to open percutaneous dilatational tracheostomy for various reasons will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
The effect of morphological structure on the percutaneous dilatational tracheostomy | April 30, 2023-October 30, 2023 (6 months)
  The relationship of anatomical position for tracheal puncture and complications with morphological structure of the patient (neck thickness, thyromental distance, thyroid cartilage measurement, cricoid cartilage measurement, jugulomental distance, distance between clavicle and cricoid cartilage)

CONTACTS AND LOCATIONS:
Overall Officials: Esin Bulut, MD, Study Director — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey
Locations (1):
- Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided